CLINICAL TRIAL: NCT06916897
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Verapamil and Food on the Pharmacokinetics of Sevasemten in Healthy Adult Subjects
Brief Title: A Study to Evaluate Effect of Verapamil and Food of Sevasemten in Healthy Volunteers
Acronym: EDG-5506-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EdgewiseTX
Record Dates: First submitted 2025-02-13; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: single dose sevasemten (Experimental): Single dose sevasemten administered on Day 1 under fasting conditions
  Interventions: Drug: sevasemten
- Treatment B: multiple doses of verapamil and single dose of sevasemten (Experimental): Multiple doses of verapamil with a single dose of sevasemten under fasting conditions
  Interventions: Drug: sevasemten; Drug: Verapamil
- Treatment C: single dose sevasemten and high-fat meal (Experimental): Single dose sevasemten under high-fat fed conditions
  Interventions: Drug: sevasemten

INTERVENTIONS:
Drug: sevasemten — single dose 10mg sevasemten administered orally
Drug: Verapamil — multiple doses 240mg verapamil
  Arms: Treatment B: multiple doses of verapamil and single dose of sevasemten

SUMMARY:
The purposes of this Phase 1 study of sevasemten are to:

1. Evaluate the effect of multiple-dose administration of verapamil on the single-dose of sevasemten in healthy adults
2. Evaluate the safety and tolerability of a single dose of sevasemten administered with and without verapamil in healthy adult subjects.
3. Evaluate the safety and tolerability of a single dose of sevasemten administered with and without food in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of non-childbearing potential)18-60 years of age, inclusive, at the screening visit.
2. Continuous non-smoker who has not used nicotine and tobacco containing products for at least 3 months prior to the first dosing based on subject self-reporting.
3. Body mass index (BMI) ≥ 18.0 and < 30.0 kg/m2 at the screening visit.
4. Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, or ECGs.
5. Willing and able to comply with the protocol.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
2. History or presence of alcohol or drug abuse (except for use of cannabis products) within the past 2 years prior to first dosing.
3. Female subjects of childbearing potential.
4. Alcohol consumption > 14 drinks per week for males or ˃ 7 drinks for females within 45 days prior to the screening visit.
5. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit.
6. Any drugs known to be moderate or strong inducers of CYP3A4 enzymes/or P glycoprotein, including St. John's Wort, beginning 28 days prior to the first dosing.
7. Is lactose intolerant.
8. Participation in another clinical study within 30 days or within 5 half-lives (if known), prior to first dosing, whichever is longer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic | Up to 46 days of monitoring
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration (AUC0-t) for sevasemten and metabolites administered with and without verapamil
Pharmacokinetic | Up to 46 days of monitoring
  The maximum observed concentration (Cmax) for sevasemten and metabolites administered with and without verapamil
Pharmacokinetic | up to 42 days of monitoring
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration (AUC0-t) for sevasemten and metabolites under fasting and fed conditions
Pharmacokinetic | up to 42 days of monitoring
  The maximum observed concentration (Cmax) for sevasemten and metabolites under fasting and fed conditions
Pharmacokinetic | up to 42 days of monitoring
  The time to reach the maximum observed concentration (Tmax) for sevasemten and metabolites under fasting and fed conditions
Pharmacokinetic | up to 42 days of monitoring
  The lag time, time delayed between drug administration and the onset of absorption (Tlag), for sevasemten and metabolites under fasting and fed conditions

SECONDARY OUTCOMES:
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of treatment emergent adverse events in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal chemistry test results in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal hematology test results in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal urinalysis test results in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal heart rate results in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal blood pressure results in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal body temperature results in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal respiratory rate results in those with a single dose of sevasemten administered with and without verapamil and with or without food
Safety and Tolerability | Up to 46 days of monitoring
  Incidence of abnormal 12-lead ECG results in those with a single dose of sevasemten administered with and without verapamil and with or without food

CONTACTS AND LOCATIONS:
Overall Officials: Roxana D Dreghici, MD, Study Chair — Edgewise Therapeutics, Inc.
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - Celerion, Lincoln, Nebraska